CLINICAL TRIAL: NCT04522115
Title: Effect of Exercise in Obese Patients With Chronic Kidney Diseases
Brief Title: Exercise for Chronic Kidney Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manal k. youssef, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T. REC/012/002608
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Chronic Kidney Failure
Keywords: chronic kidney failure; obesity; exercises
MeSH Terms: conditions — Kidney Failure, Chronic; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: group 1 received aerobic exercises and group 2 received resistance exercises.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic training (Experimental): Each exercise training session included 3 to 5 minutes of warm-up, range-of-motion exercises, interval training(aerobic training), cool-down, and post-exercise range-of-motion exercises. Patients exercise at 40 to 60% of maximum heart rate.
  Interventions: Other: exercises
- Resistance training (Experimental): Resistance exercise training of the lower extremities was performed three times per week. Starting weights for knee extension and hip abduction and flexion were determined from a three-repetition maximum (3RM) using ankle weights that can be adjusted in 1 lb. increments. A 3RM is the maximum weight that can be lifted three times with proper technique. Training started at approximately 60% of 3RM for two sets of 10 repetitions and was increased to three sets as tolerated.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Group(1) aerobic training: Each exercise training session included 3 to 5 minutes of warm-up, range-of-motion exercises, interval training(aerobic training), cool-down, and post-exercise range-of-motion exercises. Patients exercise at 40 to 60% of maximum heart rate.
  Group(2) resistance exercise: training of the lower extremities was performed three times per week. Starting weights for knee extension and hip abduction and flexion were determined from a three-repetition maximum (3RM) using ankle weights that can be adjusted in 1 lb. increments. A 3RM is the maximum weight that can be lifted three times with proper technique. Training started at approximately 60% of 3RM for two sets of 10 repetitions and was increased to three sets as tolerated.
  Other Names: resistance exercises

SUMMARY:
PURPOSE: To compare between the effect of aerobic exercise and resistance exercises on patients with obese chronic kidney diseases.

BACKGROUND: excessive adiposity is well recognized as an amplifier for the risk of renal disease progression in patients with chronic kidney diseases of various aetiology. Renal alterations induced by obesity include hyperfiltration, pathological proteinuria/ albuminuria and reduced glomerular filtration rate HYPOTHESES: There will not significantly effect of neither aerobic nor resistance on obesity, in patient with chronic kidney disease.

RESEARCH QUESTION: Aerobic exercise and resistance exercise which of them has significant effect on obesity in patient with chronic kidney disease?

DETAILED DESCRIPTION:
Questions: Does exercise improve physical performance, activity, and quality of life in obese diabetic patients with chronic kidney disease? Design: Randomized controlled trial with concealed allocation, intention-to-treat analysis, and blinded assessment.

Participants: Sixty people aged between 35and 60 years were admitted to a department of Internal medicine .Cairo University hospitals divided randomly into two Groups Intervention: group 1 received aerobic exercises. Patients exercise at 40 to 60% of maximum heart rate. The exercise period comprised the following: the warming up phase (3-5 min), which included aerobic movement exercise of range of motion joints: rotating the wrist (20 rpm clockwise and 20 rpm counter clockwise), wrist up and down (up to 20 moves on the forearm), ankle twisting motion (40 rotations clockwise and counterclockwise around the ankles), and ankles up and down (20 times); the actual phase (20-30 min), which included cycle ergo meter exercise with 12-13 rated perceived exertion; and finally the cooling down phase (3-5 min) in the form of the same aerobic movements as performed in the warming up phase. Exercises done three times per week for three months and group 2 received resistance exercises.training of the lower extremities was performed three times per week for three months. Starting weights for knee extension and hip abduction and flexion were determined from a three-repetition maximum repetition maximum(RM) using ankle weights that can be adjusted in 1 lb. increments. A RM is the maximum weight that can be lifted three times with proper technique. Training started at approximately 60% of 3 RM for two sets of 10 repetitions and was increased to three sets as tolerated. When patients could perform three sets with correct technique, the weight was increased. In addition to knee extension and hip flexion and abduction, ankle dorsiflexion and plantar flexion were performed during each exercise session Outcome measures: physical activity was measured via timed up and go test, sit to stand test, number of sit-to-stand-to-sit cycles in 60 seconds, 6 minutes walking test. Obesity was measured by BMI, waist circumference and waist to hip ratio. Also Blood pressure (systolic/diastolic blood pressures, Mean blood pressure, heart rate and blood glucose were measured before exercise. The perception of exercise intensity was assessed by Original Borg Scale. All measurements were taken at the beginning and after three months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease Stages 2-4
* body mass index ≥30
* Diabetes mellitus

Exclusion Criteria:

* Uncontrolled hypertension
* Uncontrolled diabetes mellitus.
* Cardiac failure
* Motor disorders
* Dementia

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Body mass index | 12 week
  The weight by kilogram divided by height in square meters.

CONTACTS AND LOCATIONS:
Overall Officials: Manal K Youssef, phD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2012-11-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT04522115/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04522115/SAP_001.pdf